CLINICAL TRIAL: NCT03105622
Title: Does Exercising With a Screen or Music Lead to Post-exercise Energy Compensation in Adolescents?
Brief Title: Exercising With a Screen or Music and Post-exercise Energy Compensation in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Jean-Philippe Chaput, Research Scientist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17/02X
Record Dates: First submitted 2017-03-28; First posted 2017-04-10 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Exercise; Screen; Music; Energy compensation; Adolescents; Running+screen; Running+music; Running without stimulus (control condition)
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Running+screen (Experimental): Running on a treadmill at 60% VO2peak for 30 minutes while watching television.
  Interventions: Behavioral: TV and music
- Running+music (Experimental): Running on a treadmill at 60% VO2peak for 30 minutes while listening to music.
  Interventions: Behavioral: TV and music
- Running without stimulus (control condition) (Experimental): Running on a treadmill at 60% VO2peak for 30 minutes with no other stimuli.
  Interventions: Behavioral: TV and music

INTERVENTIONS:
Behavioral: TV and music — Watching TV or listening to music while running on a treadmill

SUMMARY:
OBJECTIVE AND HYPOTHESIS:

The objective of this study will be to examine the effects of watching a screen or listening to music while exercising on acute energy intake and expenditure. It is hypothesized that the post-exercise energy compensation will be greater in both conditions with stimuli (i.e., screen and music) compared with the control condition (i.e., exercise alone).

STUDY DESIGN:

Randomized, 3-condition crossover study (within-subjects experimental design).

PARTICIPANTS:

The present study will recruit 25 male adolescents between the ages of 13 and 17 years. Participants will be recruited via advertisements and word of mouth (first come first served approach).

OVERVIEW OF THE STUDY PROTOCOL:

Preliminary Visit The participants will attend one baseline session and three experimental sessions. The preliminary visit will include measurements related to anthropometry (body weight, height, waist circumference) and resting metabolic rate. Participants will also complete questionnaires in order to better characterize them.

Experimental Sessions Each participant will be engaged in each of the following three 30-min experimental conditions followed by an ad libitum lunch: (1) walking/jogging on a treadmill at 60% of VO2 peak while watching a screen (exercise + screen); (2) walking/jogging on a treadmill at 60% of VO2 peak while listening to music (exercise + music); and (3) walking/jogging on a treadmill at 60% of VO2 peak with no other stimulus (control condition).

MEASUREMENTS:

The main measures for this study include: anthropometric measurements, food intake, appetite sensations, energy expenditure, resting metabolic rate, and ratings of perceived exertion.

OUTCOME MEASURES:

The primary outcome measure will be post-exercise energy compensation. The food intake outcome will be assessed by using an ad libitum test meal immediately after the conditions and a dietary record for the remainder of the day. The energy expenditure outcome will be assessed by using an Actical accelerometer until bedtime. The secondary outcome measures will include appetite sensations and the ratings of perceived exertion (OMNI scale).

ELIGIBILITY:
Inclusion Criteria:

- Male adolescents between 13 and 17 years

Exclusion Criteria:

* Smoking
* Unstable body weight (±4 kg) during the 3 months preceding testing
* Excessive alcohol intake (>15 drinks/week)
* Celiac disease
* Metabolic disease (e.g., thyroid disease, heart disease, diabetes)
* Medication use that could interfere with the outcome variables
* Irregular sleeping pattern (e.g., shift work or working overnight shifts)
* Iinability to comply with the protocol.

Ages: 13 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Post-exercise energy compensation (kcal/day) | Over 24 hours
  Energy balance for the remainder of the day (kcal/day)

SECONDARY OUTCOMES:
Ratings of perceived exertion | While running on the treadmill (time 0, 5, 10, 15, 20, 25, and 30 min)
  OMNI scale
Appetite sensations | 4 time points: 7:45am, 10:25am, 11:05am, and 11:30am
  Visual analogue scales (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- CHEO Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Livock H, Barnes JD, Pouliot C, LeBlanc AG, Saunders TJ, Tremblay MS, Prud'homme D, Chaput JP. Watching television or listening to music while exercising failed to affect post-exercise food intake or energy expenditure in male adolescents. Appetite. 2018 Aug 1;127:266-273. doi: 10.1016/j.appet.2018.05.016. Epub 2018 May 14. PMID 29772291

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03105622/Prot_SAP_000.pdf